CLINICAL TRIAL: NCT00344526
Title: Autologous Stem Cell Transplantation (ASCT) Versus Oral Melphalan and High-Dose Dexamethasone in Patients With AL (Primary)Amyloidosis. A Prospective Randomized Trial .
Brief Title: Intensive Versus Conventional Treatment in Patients With Primary Amyloidosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Collaborators: Ministry of Health, France (Other Government)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I00001
Record Dates: First submitted 2006-06-22; First posted 2006-06-26 (Estimated); Last update posted 2007-06-28 (Estimated); Status verified 2007-06

CONDITIONS: Primary Systemic Amyloidosis (AL)
Keywords: AL amyloidosis; Autologous stem cell transplantation; Melphalan; Dexamethasone
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — Melphalan; Dexamethasone

INTERVENTIONS:
Drug: Melphalan
Drug: Dexamethasone
Procedure: Autologous stem cell transplantation

SUMMARY:
AL amyloidosis is caused by a clonal plasma cell dyscrasia and characterized by progressive deposition of amyloid fibrils derived from monoclonal Ig light chains, leading to multisystem organ failure and death. The prognosis for AL amyloidosis with conventional treatment remains poor, Autologous stem cell transplantation (ASCT) for AL amyloidosis produces high hematologic and organ responses. However, treatment-related mortality remains high and reported series are subject to selection bias.

DETAILED DESCRIPTION:
A prospective randomized trial was conducted to compare in AL amyloidosis ASCT (melphalan 140 or 200 mg/m2 depending on age and clinical status supported with ASCT collected with G-CSF alone) and the oral regimen M-Dex (melphalan 10 mg/m2 and dexamethasone 40 mg for 4 days each months up to 18 months). The objectives were to compare survival and hematologic and clinical responses.

ELIGIBILITY:
Inclusion Criteria:

* below 70 years of age
* biopsy proven systemic AL amyloidosis
* no more than 2 prior courses of chemotherapy
* ECOG performance status < 3
* Informed written consent

Exclusion Criteria:

* localized amyloidosis
* HIV seropositivity
* previous myelodysplasia
* concomitant serious disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2000-01; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
survival

SECONDARY OUTCOMES:
hematologic responses
clinical responses

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Jaccard, MD, Principal Investigator — CH Limoges
Locations (8):
- France (8):
  - Service des Maladies du Sang, Lille
  - Service d'Hématologie et de Thérapie cellulaire, Limoges
  - Service d'hématologie clinique, Nantes
  - Service d'hématologie Clinique, Groupe Hospitalier Pitié-Salpétrière, Paris
  - Service d'hématologie clinique, Hôpital Necker, Paris
  - Service d'immuno-hématologie, Hôpital Saint-Louis, Paris
  - Service d'hématologie, Toulouse
  - Hématologie Clinique, Tours

REFERENCES:
- [Derived] Jaccard A, Moreau P, Leblond V, Leleu X, Benboubker L, Hermine O, Recher C, Asli B, Lioure B, Royer B, Jardin F, Bridoux F, Grosbois B, Jaubert J, Piette JC, Ronco P, Quet F, Cogne M, Fermand JP; Myelome Autogreffe (MAG) and Intergroupe Francophone du Myelome (IFM) Intergroup. High-dose melphalan versus melphalan plus dexamethasone for AL amyloidosis. N Engl J Med. 2007 Sep 13;357(11):1083-93. doi: 10.1056/NEJMoa070484. PMID 17855669